CLINICAL TRIAL: NCT02032615
Title: Let's Be Well Red (LBWR)
Brief Title: Let's be Well Red: Efficacy of Gudness Bars in Improving the Hemoglobin and Hematocrit Levels of Anemic Subjects
Acronym: LBWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00051046
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2015-08

CONDITIONS: Treatment and Prevention of Anemia After Administration of Gudness Nutrition Bar
Keywords: anemia
MeSH Terms: conditions — Anemia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education plus Gudness Nutritional Bar (Active Comparator): Subjects will receive education about anemia and will consume Gudness Nutrition bars for 3 months
  Interventions: Dietary Supplement: Education plus Gudness Nutritional Bar
- Education with no nutrition bar (Placebo Comparator): Subjects will receive education about anemia but will not receive nutrition bar
  Interventions: Other: Education

INTERVENTIONS:
Dietary Supplement: Education plus Gudness Nutritional Bar
  Arms: Education plus Gudness Nutritional Bar
Other: Education
  Other Names: Education about Anemia
  Arms: Education with no nutrition bar

SUMMARY:
To test the efficacy of Gudness Bars in improving the hemoglobin and hematocrit levels of anemic subjects longitudinally.

To quantify the demographics of subjects attending anemia testing camps through LBWR and to explore correlations with the demographics data.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18-35 years age

Exclusion Criteria:

* Known allergy towards nuts.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 358 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 3 months
  Measure hemoglobin levels before and after administration of Gudness nutrition bar.
Hematocrit level | 3 months
  Measure Hematocrit levels before and after administration of Gudness nutrition bar.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Clements, MD, Principal Investigator — Duke University
Locations (1):
- Lets Be Well Red, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Mehta R, Platt AC, Sun X, Desai M, Clements D, Turner EL. Efficacy of iron-supplement bars to reduce anemia in urban Indian women: a cluster-randomized controlled trial. Am J Clin Nutr. 2017 Mar;105(3):746-757. doi: 10.3945/ajcn.115.127555. Epub 2017 Jan 18. PMID 28100507